CLINICAL TRIAL: NCT03517995
Title: Randomized, Phase II Clinical Trial of Sulforaphane in Bladder Cancer Chemoprevention
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Grant not approved
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MCC-19574
Record Dates: First submitted 2018-04-26; First posted 2018-05-08 (Actual); Last update posted 2020-05-28 (Actual); Status verified 2020-02

CONDITIONS: Bladder Cancer; Bladder Tumor; Urothelial Carcinoma
Keywords: primary bladder tumor; non-muscle invasive bladder tumor; muscle invasive bladder tumor; sulforaphane; chemoprevention
MeSH Terms: conditions — Urinary Bladder Neoplasms; Carcinoma, Transitional Cell

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sulforaphane Plus Surgery (Active Comparator): Sulforaphane Administration prior to bladder cancer surgery.
  Interventions: Drug: Sulforaphane Administration; Procedure: Standard of Care Surgery
- Placebo Plus Surgery (Placebo Comparator): Placebo Administration prior to bladder cancer surgery.
  Interventions: Other: Placebo Administration; Procedure: Standard of Care Surgery

INTERVENTIONS:
Drug: Sulforaphane Administration — 1 capsule (10 mg Prostaphane) taken two times per day (2 capsules, 20 mg Prostaphane total).
  Other Names: Prostaphane
  Arms: Sulforaphane Plus Surgery
Other: Placebo Administration — 1 capsule (placebo) taken two times per day (2 capsules total).
  Arms: Placebo Plus Surgery
Procedure: Standard of Care Surgery — The study will be conducted during the time from when participants are diagnosed with bladder cancer to when they undergo a surgical procedure for the treatment or removal of their bladder cancer. The surgical procedure is done as a part of their regular medical care.
  Other Names: post study treatment surgery; bladder cancer surgery

SUMMARY:
The main purpose of this study is to see if Prostaphane is effective and can help reduce the progression of bladder cancer. Researchers also want to find out if Prostaphane is safe and tolerable, and to evaluate how Prostaphane works to reduce the progression of bladder cancer. This study will compare Prostaphane with a placebo to see if taking Prostaphane is better than taking a placebo. A placebo is a pill that looks like Prostaphane but has no drug or other active ingredients in it.

The study will be presented to eligible patients by the patient's surgeon at the time when an appointment is made for cystoscopy for suspicion of bladder cancer (BC) or to confirm BC diagnosis.

DETAILED DESCRIPTION:
The study will be presented to eligible patients by the patient's surgeon at the time when an appointment is made for cystoscopy for suspicion of bladder cancer (BC) or to confirm BC diagnosis.

Participants will be asked to spend 21 to 30 days in this study. The study will be conducted during the time from when the participant is diagnosed with bladder cancer to when they undergo a surgical procedure for the treatment or removal of their bladder cancer. The surgical procedure is done as a part of their regular medical care. Participants will be asked to come for 1 additional visit as part of this research study at the midpoint between their biopsy and surgery.

ELIGIBILITY:
Inclusion Criteria:

* Men and women; age ≥18 years; evidence of non-muscle invasive or muscle invasive primary bladder tumor (urothelial carcinoma +/- variant histology) discovered on cystoscopy or radiologic imaging performed within 60 days of randomization; with no evidence of distant metastases; planned Transurethral Resection+B21 (TURBT), cystoscopy with biopsies or cystectomy (total or partial);
* Absent prior pelvic radiation; normal organ function;
* Absent neoadjuvant chemotherapy (refusal or ineligibility); (the participant may have prior intravesical treatment exposure (including Bacillus Calmette-Guerin (BCG), mitomycin, gemcitabine, valrubicin, docetaxel, etc.) for bladder cancer (BC) (excluding primary bladder radiation therapy) provided that treatment was completed greater than 30 days prior to the patient's randomization visit);
* Non-smokers (urinary cotinine tested);
* Agree to restrict dietary sources of Sulforaphane (SFN) to 3 or 5 servings/week and abstain from consuming SFN supplements beginning three days prior to start of study and throughout duration of the study;
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2;
* Willing to discontinue current vitamin/mineral supplement use and substitute with a standard multivitamin supplement provided for the study;
* Willing to use an effective method of contraception, if the partner is of child-bearing age, while on study;
* Willing to comply with proposed visit and treatment schedule;
* Able to understand and willing to sign a written informed consent document;
* Participants must have normal organ and marrow function.

Exclusion Criteria:

* Evidence of other cancers (excluding non-melanoma skin cancer) or metastatic disease;
* Prior pelvic radiation; concurrent systemic chemotherapy for any other cancer, excluding non-melanoma skin cancer;
* Any treatment for the bladder tumor other than intravesical therapy;
* Prior treatment with a known histone deacetylase inhibitor (including but not limited to valproic acid, suberoylanilide hydroxamic acid (SAHA), Panobinostat (LBH589), etc.) within 6 months prior to starting study treatment or while on study therapy;
* Current treatment with warfarin;
* Use of dietary supplements or herbal remedies which may affect the study outcome - unless the participant is willing to discontinue taking them for 1 month prior to starting study;
* Usual consumption of > 5 servings per week of brassica vegetables;
* Gastrointestinal ailments which would interfere with the ability to adequately absorb SFN;
* Allergy/known intolerance to cruciferous vegetables;
* Used antibiotics (more than 3 doses) within 10 days prior to study (day -14 prior to study randomization);
* Current smoker.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-04 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Magnitude of Change | Up to 30 days
  Magnitude of change in Intermediate Endpoint Biomarkers (IEBs) of proliferation (Ki-67 expressing cells- an independent marker of poor prognosis in bladder cancer (BC)) from baseline to end of treatment with 20 mgs Prostaphane® [Nutinov Labs, France] containing 200 μmol of Sulforaphane (SFN) a day at 3-4 weeks (maximum 30 days) in BC cells and benign/adjacent cells.

SECONDARY OUTCOMES:
Effectiveness of Sulforaphane vs. Placebo | End of study, approximately 30 days
  Effectiveness of SFN at this dose (vs. placebo) as indicated by modulation of other IEBs of proliferation, apoptosis and phase II enzymes, as well as the potential molecular mechanism of SFN, we will measure changes in: (i) BC histology grade; (ii) labeling index of a sensitive biomarker that is a member of DNA replication origin licensing complex, Mcm2; (iii) apoptosis (Caspase-3); (iv) Phase II enzymes (glutathione transferases, epoxide hydrolase, Nicotinamide adenine dinucleotide phosphate (NAD(P)H): quinone reductase, and glucuronosyltransferases); (v) Nrf2 and Transcription factor (NF-kB) signaling, from baseline to end of treatment in BC cells and benign/adjacent cells.
Occurrence of Adverse Events per Study Arm | End of study, approximately 30 days
  Safety of SFN at this dose (vs. Placebo) as indicated by incidence of adverse events and toxicities, monitored using Common Toxicity Criteria version 5.0, complete blood count (CBC), and complete metabolic panel (CMP) from baseline at mid-point and at end of trial.
Mid-study Bioavailability of Sulforaphane | Mid-study, approximately 15 days
  Bioavailability, of SFN at this dose vs. Placebo. Investigators will measure change in SFN in plasma and bladder tissue from baseline, at mid-point and at end of study.
End of Study Bioavailability of Sulforaphane | End of study, approximately 30 days
  Bioavailability, of SFN at this dose vs. Placebo. Investigators will measure change in SFN in plasma and bladder tissue from baseline, at mid-point and at end of study.
Adherence of Sulforaphane vs. Placebo | End of study, approximately 30 days
  Adherence based on pill counts and diet and pill logs from baseline.
Acceptability of Sulforaphane vs. Placebo | End of study, approximately 30 days
  Acceptability based on pill counts and diet and pill logs from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Nagi Kumar, Ph.D, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (2):
- United States (2):
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - James A. Haley Veteran's Administration Hospital, Tampa, Florida